CLINICAL TRIAL: NCT02600793
Title: Ceftaroline Diffusion Into Cerebrospinal Fluid of Children With Ventriculitis Due to Ventriculoperitoneal Shunt (VPS) Infection
Brief Title: Ceftaroline Diffusion Into Cerebrospinal Fluid of Children
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Basim Asmar (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor-Investigator, Basim Asmar, Professor of Pediatrics, Wayne State University
Organization: Wayne State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CeftarolineCSF2013
Record Dates: First submitted 2015-11-06; First posted 2015-11-09 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Cerebrospinal Fluid Shunts; Ventriculoperitoneal Shunt
MeSH Terms: interventions — Ceftaroline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Single dose IV ceftaroline will be administered
  Interventions: Drug: Ceftaroline

INTERVENTIONS:
Drug: Ceftaroline — Following Ceftaroline single IV dose, 3 blood and cerbrospinal fluid samples will be collected
  Other Names: Ceftaroline Fosamil; Teflaro

SUMMARY:
Ceftaroline fosamil is an intravenous (IV) drug that belongs to a group of antibiotics called cephalosporins . Antibiotics are drugs used to treat infections. Clinical studies in adults patient shave shown ceftaroline fosamil to be effective against many bacteria that are resistant to other currently approved antibiotics. Some of these bacteria may be responsible for infections in the central nervous system.The main aim of this study is to gather information to determine how much of a single IV dose of ceftaroline fosamil will enter into a child's CSF so that the benefit of giving ceftaroline fosamil to children with infections can be better determined.

DETAILED DESCRIPTION:
Children 6 months to 17 years of age admitted to the hospital because of infected VPS (ventriculitis) will be eligible for the study. A total of twelve eligible patients will be included in the study. Eligible study subjects would be patients who have undergone VPS removal and placement of EVD tubing and are being treated with standard IV antibiotics for ventriculitis. CSF cultures are obtained before antibiotics treatment is initiated. Standard initial antibiotics regimen is usually IV ceftriaxone and vancomycin. The antibiotics regimen is subsequently adjusted based on the pathogen recovered from the CSF culture. Total IV antibiotic treatment is usually 14 days. Following clearance of the infection the patient undergoes new VPS insertion by neurosurgery service.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months - 17 years
* Ventriculitis due to VPS infection (abnormal CSF parameters consistent with meningeal inflammation and/or positive CSF culture)
* VPS is externalized and External Ventriculostomy Drain (EVD) is in place
* Patient has IV access and is receiving antibiotic treatment for VPS infection
* Parent/Guardian signed written informed consent
* Negative urine or serum pregnancy test for females of child-bearing potential

Exclusion Criteria:

* Known Allergy to beta-lactam antibiotics
* Moderate to severe renal impairment (Creatinine clearance < 50mL/minute)
* Parent/Guardian written consent cannot be obtained
* Positive urine or serum pregnancy test

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic assessment of Ceftaroline diffusion from blood into the Cerbrospinal fluid. | 8 hours
  Serial collection of three blood and three cerbrospinal fluid sample over 8 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Michigan, Detroit, Michigan, United States